CLINICAL TRIAL: NCT00324051
Title: PREFERENCE: 12-Week Open Label Trial On Olanzapine Orodispersible Tablet Vs. Oral Olanzapine Preference Study
Brief Title: Patient's Preference Between Conventional Oral Olanzapine Tablet vs Olanzapine Orodispersible Tablet
Acronym: PREFERENCE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 10960; F1D-VI-S067 (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-05-08; First posted 2006-05-10 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: olanzapine therapy

SUMMARY:
The purpose of the study is to estimate drug preference of stable schizophrenic patients who will be treated with olanzapine orodispersible tablets for 6 weeks then with olanzapine tablets for 6 weeks and vice-versa.

ELIGIBILITY:
Inclusion Criteria:

* You are an outpatient diagnosed with stable schizophrenia.
* You are a male or female in the age of 18 to 65 years old.
* You are retrospectively judged by investigators, based on clinical interview and impression, to have been stable for at least 4 weeks.
* You must be able to take olanzapine orodispersible in a single daily dose.
* You are treated with conventional oral olanzapine tablet (as monotherapy) for at least 1 month.

Exclusion Criteria:

* You have used olanzapine in the past and are no longer using it because of a bad reaction.
* You have known Human immunodeficiency virus positive (HIV+) status.
* You have known uncorrected, narrow angle glaucoma.
* You have known Leukopenia, (abnormally low white blood cell count).
* You have a serious or uncontrolled illness (for example: liver disease, history of heart disease, or inadequately controlled diabetes.)
* You have Parkinson's disease.
* You are a female patient who is either pregnant or nursing
* You are taking medications that are not allowed in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2006-05; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Patient preference measured by a simple preference question.

SECONDARY OUTCOMES:
Better treatment adherence as measured by DAI-10
Safety and tolerability as measured by AMDP-5
Determine the predictors of drug compliance
Mean change from baseline to endpoint in body mass index (BMI)
Compare serum ghrelin levels
Differences in subjective appetite from baseline to endpoint using a visual analog scale (VAS)
Effect on the medication compliance, level of medication supervision, and willingness to remain on medication, as measured by Medication Adherence Form (MAF)
Patient preference of the paranoid sub population as measured by a simple preference question

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (8):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio de Janeiro, Brazil
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Constanța, Romania
- Turkey (Türkiye) (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Adana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ankara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bursa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elâzığ
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gaziantep
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Istanbul

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Result] Bitter I, Treuer T, Dilbaz N, Oyffe I, Ciorabai EM, Gonzalez SL, Ruschel S, Salburg J, Dyachkova Y. Patients' preference for olanzapine orodispersible tablet compared with conventional oral tablet in a multinational, randomized, crossover study. World J Biol Psychiatry. 2010 Oct;11(7):894-903. doi: 10.3109/15622975.2010.505663. PMID 20653494
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com